CLINICAL TRIAL: NCT03548909
Title: VITROS Immunodiagnostic Products NT-proBNP II
Status: Completed | Type: Observational
Sponsor: Ortho-Clinical Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-001
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
Keywords: NT-proBNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Lithium Heparin, and EDTA
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- ED Setting: An acute HF population enrolled at EDs. Testing of clinical samples will be performed with the VITROS Immunodiagnostic Products NT-proBNP II assay.
  Interventions: Diagnostic Test: VITROS Immunodiagnostic Products
- Outpatient Setting: A non-acute population enrolled at outpatient centers.Testing of clinical samples will be performed with the VITROS Immunodiagnostic Products NT-proBNP II assay.
  Interventions: Diagnostic Test: VITROS Immunodiagnostic Products

INTERVENTIONS:
Diagnostic Test: VITROS Immunodiagnostic Products — NT-proBNP II assay

SUMMARY:
Amino Terminal pro-Brain Natriuretic Peptide (NTproBNP) is secreted in conditions of cardiac wall stress. NTproBNP levels are used in addition to clinical assessment to diagnose heart failure (HF). The purpose of this clinical study is to collect data to substantiate the use of the VITROS NT-proBNP II assay.

DETAILED DESCRIPTION:
A prospective clinical sample collection and NT-proBNP testing will be conducted in two populations. Patients presenting to the Emergency Department (ED) and patients presenting to outpatient centers will be approached for enrollment.

Clinical and laboratory data will be collected to demonstrate product performance compared to adjudicated clinical diagnosis. Approximately 4300 evaluable subjects at geographically dispersed sites in the US will be enrolled in the study.

Sample collection and testing of clinical samples with the VITROS NT-proBNP II assay will be performed under two separate protocols.

ELIGIBILITY:
Acute HF Population (ED setting):

Inclusion Criteria:

* Subjects must have suspicion of HF and acute symptoms at presentation.
* Subjects must be at least 22 years of age.
* Subjects must be willing and able to provide informed consent.

Exclusion Criteria:

* Acute symptoms clearly not secondary to HF.
* Subjects with renal disease on dialysis.
* Subjects unable to comply with the study requirements.

Population with suspicion of HF (Outpatient Setting):

Inclusion Criteria:

* Subjects must be at least 22 years of age.
* Subjects must be willing and able to provide informed consent.
* Subjects who present to outpatient centers with suspicion HF.

Exclusion Criteria:

* Symptoms clearly not secondary to HF.
* Subjects with renal disease on dialysis.
* Subjects unable to comply with the study requirements.
* Subjects previously diagnosed with heart failure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The ED population represents an acute HF population enrolled at Emergency Departments. Patients presenting with a suspicion of HF and acute symptoms will be approached for enrollment.
  The outpatient population represents a population with suspicion of HF presenting to outpatient centers. Patients presenting with a suspicion of HF will be approached for enrollment.
Sampling Method: Probability Sample
Enrollment: 3246 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the VITROS NT-proBNP II assay | Single blood draw upon study entry 1day
  Establish the performance of the VITROS NT-proBNP II assay against the adjudicated diagnosis.

SECONDARY OUTCOMES:
Heart Failure Severity Assessment | Single blood draw upon study entry 1 day
  Demonstrate that the VITROS NT-proBNP II assay may be used for assessment of heart failure severity.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Christenson, PhD, Principal Investigator — University of Maryland, College Park
Locations (25):
- United States (25):
  - Drug Research Analysis Corp, Montgomery, Alabama
  - University of Arizona Banner - University Medical Center South Campus, Tucson, Arizona
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - University of California Davis Health, Sacramento, California
  - University of California San Diego Health, San Diego, California
  - Northwestern University, Evanston, Illinois
  - Indiana University Health Hospital (Eskenazi & Methodist), Indianapolis, Indiana
  - Southern Clinical Research, Zachary, Louisiana
  - University of Maryland (Baltimore & St. Joseph), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State University (Harper), Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital (Royal Oak & Troy), Royal Oak, Michigan
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - Charlotte-Mecklenburg Hospital Authority (Carolinas Healthcare System), Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine (Ben Taub), Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - INOVA Healthcare Services, Falls Church, Virginia

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Richards AM, Nicholls MG, Yandle TG, Frampton C, Espiner EA, Turner JG, Buttimore RC, Lainchbury JG, Elliott JM, Ikram H, Crozier IG, Smyth DW. Plasma N-terminal pro-brain natriuretic peptide and adrenomedullin: new neurohormonal predictors of left ventricular function and prognosis after myocardial infarction. Circulation. 1998 May 19;97(19):1921-9. doi: 10.1161/01.cir.97.19.1921. PMID 9609085
- [Background] Valli N, Gobinet A, Bordenave L. Review of 10 years of the clinical use of brain natriuretic peptide in cardiology. J Lab Clin Med. 1999 Nov;134(5):437-44. doi: 10.1016/s0022-2143(99)90163-4. PMID 10560935
- [Background] Darbar D, Davidson NC, Gillespie N, Choy AM, Lang CC, Shyr Y, McNeill GP, Pringle TH, Struthers AD. Diagnostic value of B-type natriuretic peptide concentrations in patients with acute myocardial infarction. Am J Cardiol. 1996 Aug 1;78(3):284-7. doi: 10.1016/s0002-9149(96)00278-0. PMID 8759805
- [Background] McDonagh TA, Robb SD, Murdoch DR, Morton JJ, Ford I, Morrison CE, Tunstall-Pedoe H, McMurray JJ, Dargie HJ. Biochemical detection of left-ventricular systolic dysfunction. Lancet. 1998 Jan 3;351(9095):9-13. doi: 10.1016/s0140-6736(97)03034-1. PMID 9433422
- [Derived] Daniels LB, Ajongwen P, Christenson RH, Clark CL, Diercks DB, Fermann GJ, Mace SE, Mahler SA, Pang PS, Rafique Z, Runyon MS, Tauras J, deFilippi CR. Clinical Performance of an N-Terminal Pro-B-Type Natriuretic Peptide Assay in Acute Heart Failure Diagnosis. J Appl Lab Med. 2025 Mar 3;10(2):325-338. doi: 10.1093/jalm/jfae107. PMID 39495056